CLINICAL TRIAL: NCT05749003
Title: Effect of Sensorimotor Training Exercise After Lower Extremity Burns, Prospective Randomized Controlled Trial
Brief Title: Sensorimotor Training Exercise After Lower Extremity Burns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Morgan Allam, Assistant Professor of physical therapy for surgery, Faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004323
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2023-02

CONDITIONS: Lower Extremity Burns
Keywords: Sensorimotor training; Stability; Mobility; Balance; Burn
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sensorimotor training program group (Experimental): participants will receive Sensorimotor training exercise plus conventional physical therapy program of exercise.
  Interventions: Other: sensorimotor training exercise; Other: conventional physical therapy program of exercise.
- Control group (Other): participants will receive conventional physical therapy program of exercise.
  Interventions: Other: conventional physical therapy program of exercise.

INTERVENTIONS:
Other: sensorimotor training exercise — Patients will be trained through three stages: static, dynamic and functional. Each exercise will be repeated 3-5 times during a session and with enough periods of rest between each set of exercises. The exercise graduated from easy to more difficult and the patient was not progressed to a more difficult stage until performing the easier one.
  Arms: sensorimotor training program group
Other: conventional physical therapy program of exercise. — stretching exercise for 30 minutes, then strengthening exercise and usual burn care for the lower extremity. Exercises will be applied for 3 times a week for 8 consecutive weeks.

SUMMARY:
Burn injury affects dermal tissue which contains sensory neurones that contribute to the conscious and automatic feedback systems which in turn, control balance and coordination. Impediments arising from lower limb burn injuries are similar to those observed in other populations suffering lower limb disease or pathology and further, these complications cause balance dysfunction. Balance and mobility are complex bodily functions integral to discharge disposition, social function and quality of life. Therefore, to guide recovery accurately and facilitate rehabilitation after LLBI, multi-factorial assessment is required.

DETAILED DESCRIPTION:
Burns to the lower limbs can cause pain, scar tissue contracture, impaired sensation, muscle weakness and postural imbalance are all potential complications of lower limb burn injury (LLBI) which negatively influence a person's ability to function normally

Sensorimotor training is a special form of proprioceptive and balance exercise that was designed for management of patients with chronic musculoskeletal pain syndromes. It is based on the concept that instead of emphasizing the isolated strength of a group of muscles around a joint, we should realize the importance of the central nervous system in regulating movement in order to reach proper firing patterns for maintaining joint stability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of thermal burn injuries at the lower extremities.
* Total body surface area burned approximately from 40 to 50%.
* Patients age: 20 to 50 years.

Exclusion Criteria:

* Cognitive or mentality dysfunctions.
* Psychiatric conditions.
* Fractures.
* Pregnancy.
* Cancer.
* Severe vascular complications.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Stability assessment | 2 months
  Biodex balance scale (Biodex medical systems Inc, Shirley, New York, USA), will be used for balance assessment. Anteroposterior stability index, mediolateral stability index, and overall stability index will be used to assess fluctuations around the zero point representing standard deviations rather than around a group mean.
Balance assessment | 2 months
  The Berg balance scale includes 14 items with scores from 0 to 4. A score of 0 represents the inability to do the task, while a score of 4 represents the ability to do the task completely, according to the assigned criteria, with 56 indicates the total score.

SECONDARY OUTCOMES:
Mobility assessment | 2 months
  For assessment of mobility, the timed-up and go test was used. The test asks the participant to raise up from the sitting position followed by walking for 3 m, turning around, sitting again on the chair with his back supported, and resting his arms on the armrests. A stopwatch was used to measure the time in seconds for each participant to finish the task. The test was repeated for three trials, and the best or lowest trial time was documented for analysis.
Quality of life (36-Item Short Form Health Survey (SF-36). | 2 months
  HRQoL using the Medical Outcomes Study 36-Item Short Form Health Survey (SF-36). The SF-36 is a generic measure of HRQoL that contains 36 items grouped into: physical functioning, physical role functioning, bodily pain, general health perceptions, vitality, social role functioning, emotional role functioning, and mental health. Scores on each subscale range from 0 to 100, with 0 corresponding to the worst health status and 100 to the best health status.
Muscle Torque assessment | 2 months
  The therapist will perform the initial evaluation of knee extensor muscles of the dominant burned limb with Biodex isokinetic dynamometer (Biodex Medical System, Shiley, NY, USA, linked to IBM PC-computer software). After a 5-min warm-up on the treadmill without resistance, the participants will be positioned in an isokinetic dynamometer with hip angle of 100°. The trunk, pelvis and thigh will be stabilized using straps, in accordance with the Test and Rehabilitation System User's Guide of Biodex.

CONTACTS AND LOCATIONS:
Overall Officials: Hadaya M Eladl, PhD, Study Chair — Assisstant professor of physical therapy for surgery, Faculty of physical therapy
Locations (1):
- Nesma Morgan Allam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study results
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: Study protocol